CLINICAL TRIAL: NCT06589830
Title: A Phase 2 Study to Evaluate TL938 Combined With Trastuzumab in Patients With HER2-positive Metastatic Colorectal Cancer
Brief Title: TL938 and Trastuzumab for Patients With HER2-positive Metastatic Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Teligene Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TL-HER-202301
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer Metastatic; Advanced Colorectal Cancer
Keywords: Oncology; TL938; Colorectal Cancer; HER2
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TL938-Trastuzumab combination (Experimental): TL938-Trastuzumab combination receives TL938 capsules by mouth once daily. Trastuzumab given intravenously on Day 1 of each Cycle. Cycle length is 21 days
  Interventions: Drug: TL938 Capsules; Drug: Trastuzumab
- TL938 (Experimental): TL938 monotherapy receives TL938 capsules by mouth once daily. Cycle length is 21 days.
  Interventions: Drug: TL938 Capsules

INTERVENTIONS:
Drug: TL938 Capsules — Oral administration
Drug: Trastuzumab — Intravenous (IV) infusion
  Arms: TL938-Trastuzumab combination

SUMMARY:
This is a Phase II trial designed to determine the optimal dose and evaluate the effectiveness of TL938 and trastuzumab in treating patients with HER2+ colorectal cancer that has metastasized or recurred and is inoperable.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years old and above, male or female;
2. Her2-positive, RAS wild-type, unresectable or metastatic colorectal cancer and prior treatment with fluoropyrimidine, oxaliplatin, irinotecan, and an anti-vascular endothelial growth factor (VEGF) monoclonal antibody (mAb). Patients whose tumors were deficient in mismatch repair (dMMR) proteins or were microsatellite instability-high (MSI-H) must also have received an ant-programmed cell death protain-1 mAb;
3. At least one measurable lesion;
4. Eastern Cooperative Oncology Group (ECOG) score of 0, 1, or 2;
5. A minimum life expectancy of >3 months;
6. Adequate bone marrow reserve, hepatic, renal, and coagulation function;
7. Other inclusion criteria apply for participating in the Study. -

Exclusion Criteria:

1. Prior anti-HER2 targeting therapy;
2. Any systemic ant-tumor therapy such as chemotherapy and radiation therapy (including curative radiotherapy or spinal radiotherapy portion >30%) used within 3 weeks prior to enrollment; immunotherapy within 4 weeks; any palliative radiotherapy for nan-target lesions used to relieve symptoms within 2 weeks prior to enrollment;
3. Participation in another interventional clinical trial 2 weeks prior to enrollment or within 5haIf-lives from the last dose of IP (whichever is shorter);
4. Surgical operation (excluding aspiration biopsy) of main organs or a significant injury within 4 weeks prior to enrollment;
5. Any unresolved toxicities from prior therapy greater than Grada 1, at the time of screening;
6. Active central nervous system (CNS) metastases. Asymptomatic CNS metastases with no steroid use within the last 30 days prior to enrollment is eligible;
7. Any other primary malignant tumors within 3 years (except for cured skin basal cell carcinoma and carcinoma in situ of cervix, low risk cancer such as low grade prostate cancer or ductal carcinoma in situ of the breast;
8. Any active infection which has not been controlled at screening;
9. Other exclusion criteria apply for participating in the Study. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity, maximum tolerated dose, and recommended phase 2 dose | Pre-dose up to approximately 24 months post-dose
Objective Response Rate (ORR) by IRC | Pre-dose up to approximately 24 months post-dose

SECONDARY OUTCOMES:
Objective Response Rate (ORR) by Investigator | Pre-dose up to approximately 24 months post-dose
Duration of Response (DoR) | Pre-dose up to approximately 24 months post-dose
Disease Control Rate (DCR) | Pre-dose up to approximately 24 months post-dose
Progression Free Survival (PFS) | Pre-dose up to approximately 24 months post-dose
Time to Tumor Progression (TTP) | Pre-dose up to approximately 24 months post-dose
Time to Treatment Failure (TTF) | Pre-dose up to approximately 24 months post-dose
Time to Response (TTR) | Pre-dose up to approximately 24 months post-dose
Overall Survival (OS) | Pre-dose up to approximately 24 months post-dose
1-year Progression Free Survival | Pre-dose up to approximately 24 months post-dose
1-year Survival | Pre-dose up to approximately 24 months post-dose
Number of Participants Experiencing Adverse Events (AE) | Pre-dose up to approximately 24 months post-dose
Number of Participants Experiencing Adverse Drug Reactions (ADR) | Pre-dose up to approximately 24 months post-dose
Number of Participants Experiencing Serious Adverse Events (SAE) | Pre-dose up to approximately 24 months post-dose
Number of Participants Experiencing Serious Adverse Reactions (SAR) | Pre-dose up to approximately 24 months post-dose
Area Under The Curve (AUC) of TL938 | Pre-dose up to 24 hours post-dose
Maximum Plasma Concentration (Cmax) of TL938 | Pre-dose up to 24 hours post-dose
Minimum Plasma Concentration (Cmin) of TL938 | Pre-dose up to 24 hours post-dose
Time to Peak Drug Concentration (Tmax) of TL938 | Pre-dose up to 24 hours post-dose
TL938 half-life (T1/2) | Pre-dose up to 24 hours post-dose
Volume of Distribution (Vz/F) of TL938 | Pre-dose up to 24 hours post-dose
Apparent Clearance (CL/f) of TL938 | Pre-dose up to 24 hours post-dose

IPD SHARING:
Plan to Share IPD: No